CLINICAL TRIAL: NCT03801629
Title: Imaging the Neuroimmune Effects of Acute Opioid Administration
Brief Title: Neuroimmune Effects of Opioid Administration
Acronym: NOA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Principal Investigator, Eric Woodcock, Associate Research Scientist, Yale University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2000024785
Record Dates: First submitted 2019-01-08; First posted 2019-01-11 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Drug Effect
Keywords: Neuroimmune System; Morphine; PET Imaging; TSPO
MeSH Terms: interventions — Contraceptives, Oral

STUDY DESIGN:
Intervention Model Description: Subjects will receive a single intramuscular morphine dose: 'High' (0.07mg/kg i.m.) vs. 'Low' (0.04mg/kg i.m.)
Who Masked: Participant
Masking Description: Subjects are informed that they will receive a single morphine injection. Subjects are blinded to the morphine dose condition. Investigators and assessors are not blinded to morphine dose condition.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- High Morphine Dose (Experimental): Subjects in this experimental arm will receive a single intramuscular morphine dose (non-dominant deltoid muscle; 0.07 mg/kg).
  Interventions: Drug: High Morphine Dose
- Low Morphine Dose (Experimental): Subjects in this experimental arm will receive a single intramuscular morphine dose (non-dominant deltoid muscle; 0.04 mg/kg).
  Interventions: Drug: Low Morphine Dose

INTERVENTIONS:
Drug: High Morphine Dose — Subjects will receive an intramuscular morphine injection (0.07mg/kg) in the non-dominant deltoid muscle. Metoclopramide (10mg; oral) will be administered PRN to reduce nausea.
  Other Names: High Dose
  Arms: High Morphine Dose
Drug: Low Morphine Dose — Subjects will receive an intramuscular morphine injection (0.04mg/kg) in the non-dominant deltoid muscle. Metoclopramide (10mg; oral) will be administered PRN to reduce nausea.
  Other Names: Low Dose
  Arms: Low Morphine Dose

SUMMARY:
Preclinical research indicates acute opioid administration evokes an immune response in the periphery and brain. Here, we will translate those preclinical findings to healthy human volunteers and quantify the neuroimmune response to a morphine challenge using positron emission tomography (PET) imaging with [11C]PBR28.

DETAILED DESCRIPTION:
Subjects will be recruited from the local community via media advertisements, flyers, and word-of-mouth. Interested individuals will undergo a phone screen and in-person medical and psychiatric examination. Up to 20 eligible individuals (see Inclusion/Exclusion criteria) will be invited to participate in this study.

In a single day, subjects will complete behavioral and physiological testing, a [11C]PBR28 PET scan, and report subjective drug effects before and after a morphine challenge. Subjects will complete either a 'High' or 'Low' morphine dose condition (single-blind): 0.07mg/kg i.m. vs. 0.04mg/kg i.m., respectively. To measure the neuroimmune response to morphine, we will use [11C]PBR28 PET imaging (120-minute scans on a High Resolution Research Tomograph with Vicra motion correction). [11C]PBR28 binds with high affinity and specificity to the 18kDa translocator protein (TSPO), which is highly expressed in microglia and has been shown to respond to inflammatory challenges. TSPO volumes of distribution (VT), i.e., TSPO availability, will be quantified in brain regions of interest using multilinear analysis-1 (MA-1) with the metabolite-corrected arterial input function. The post-morphine [11C]PBR28 PET scan will occur 2-hours after the morphine challenge.

Specific Aim 1: To determine whether an acute morphine administration increases brain TSPO availability in healthy volunteers.

Hypothesis 1: Relative to pre-morphine levels, morphine will significantly increase TSPO availability across brain regions of interest, consistent with a neuroimmune response.

Specific Aim 2: To determine whether morphine evokes a dose-dependent increase in brain TSPO availability in healthy volunteers.

Hypothesis 2: Relative to pre-morphine levels, morphine will dose-dependently increase TSPO availability across brain regions of interest.

Specific Aim 3: To determine whether morphine administration increases peripheral markers of inflammation, e.g., cytokine/chemokine concentration in plasma.

Hypothesis 3: Relative to pre-morphine levels, morphine will increase cytokine/chemokine concentrations in plasma, including IL-1B, IL-2, IL-6, IL-10, TNF-a, IFNy, MCP-1, and GM-CSF, consistent with a peripheral immune response. Exploratory Hypotheses: 1) IL-1B, IL-6, TNF-a, IFNy, MCP-1, and GM-CSF will exhibit morphine dose-dependent increases in plasma. 2) The change in IL-6, TNF-a, IFN-y, and GM-CSF levels will be positively correlated with the change in brain TSPO VT levels.

Specific Aim 4: To determine whether morphine administration alters pain sensitivity, pain tolerance, cognitive function, and reward responsiveness.

Hypothesis 4: Relative to pre-morphine levels, morphine will enhance pain tolerance and impair verbal learning/memory proficiency and impair reward responsiveness. Morphine will not alter pain sensitivity, visual attention, psychomotor processing speed, or working memory proficiency. Exploratory hypotheses: 1) The change in TSPO availability in thalamus will be positively correlated with the change in pain tolerance. 2) The change in TSPO availability in hippocampus will be inversely correlated with the change in verbal learning/memory proficiency. 3) The change in TSPO availability in caudate, ACC, and OFC will be inversely correlated with the change in reward responsiveness.

Specific Aim 5: To determine whether morphine administration alters vital signs.

Hypothesis 5: Relative to pre-morphine levels, morphine will dose-dependently reduce systolic and diastolic blood pressure. Relative to pre-morphine levels, morphine will lower heart rate.

Specific Aim 6: To measure the subjective response to morphine administration.

Hypothesis 6: Relative to pre-morphine levels, morphine will dose-dependently increase subjective ratings of 'high', 'good drug effect', 'nausea', and 'bad drug effect'. Exploratory hypotheses: 1) The change in TSPO availability in caudate, ACC, and OFC will be positively correlated with the change in 'high' and 'good drug effect'. 2) The change in TSPO availability in the insula and thalamus will be positively correlated with the change in 'nausea' and 'bad drug effect'.

Specific Aim 7: To determine whether morphine administration alters peripheral stress markers of the autonomic nervous system and HPA-axis.

Hypothesis 7: Relative to pre-morphine levels, morphine will dose-dependently increase plasma levels of epinephrine, norepinephrine, and cortisol.

Specific Aim 8: To determine whether morphine administration alters peripheral markers of neurosteroids.

Hypothesis 8: Relative to pre-morphine levels, morphine will dose-dependently increase plasma levels of allopregnanolone and pregnenolone.

Specific Aim 9: To determine whether morphine administration alters peripheral markers of the metabolic hormone ghrelin.

Hypothesis 9: Relative to pre-morphine levels, morphine will dose-dependently increase plasma levels of ghrelin.

ELIGIBILITY:
PBR_Morphine Study

Inclusion Criteria:

1. Men and women aged between 21 and 50 years (driver's license or valid state ID).
2. Physically healthy by medical history, physical, neurological, EKG and laboratory examinations (reviewed by the Study Physician).
3. Normal weight, as indicated by a body mass index (BMI) and body weight ≤ 250lbs.
4. Read, comprehend, and write English at a sufficient level to complete study-related materials.
5. Able to provide voluntary and written informed consent.
6. Eligibility and willingness to participate in study procedures, including MRI and PET scanning.
7. Previous medical use of opioids without adverse reactions (≥2 lifetime uses).
8. Medically eligible to receive up to 0.1 mg/kg deltoid intramuscular morphine (based on medical history, medical exams, and not meeting any exclusion criteria below).
9. Medically eligible to receive 10mg of oral metoclopramide based on medical history, medical exams, and current medications.

Exclusion criteria:

1. Any DSM-5 Axis I disorder diagnosis based on Structured Clinical Interview for DSM-5 (SCID-5), including meeting criteria for substance dependence.
2. Any current psychotropic medication use, including MAOI use within the past 14 days
3. Recent (past 6 months) medical or non-medical opioid-use.
4. Prior medical use prescription opioids for >14 consecutive days (self-report)
5. Prior non-medical use of any opioid (i.e., recreational opioid use will be excluded).
6. Positive result on a urine drug screen (excluding marijuana).
7. Current or previous chronic pain disorder (>6 months of continuous pain).
8. 'Low affinity binding' individuals based on rs6971 polymorphism (<10% of the population).
9. For females, pregnancy (positive urine test).
10. Current use of non-steroidal anti-inflammatory medications or statins.
11. Medical contraindication to receive up to 0.1 mg/kg intramuscular morphine administration as determined by Study Physician. This includes:

    1. known hypersensitivity/allergy to morphine;
    2. acute or severe bronchial asthma;
    3. known or suspected gastrointestinal obstruction, including paralytic ileus;
    4. seizure disorder;
    5. concomitant use of a benzodiazepine or any other CNS depressant;
    6. any other significant medical condition, that in the opinion of the Study Physician and Investigators, could: put the patient at risk because of participation in the study, or influence the results of the study, or cause concern about the patient's ability to successfully complete in the study.
12. Known family history (first-degree relative) of opioid-use disorder or alcohol-use disorder.
13. MRI contraindications, including metal in body (or work in metal/machine shop), pacemaker, claustrophobia, or inability to tolerate MRI scanning.
14. Medical contraindications to metoclopramide, as determined by the Study Physician, including:

    1. known hypersensitivity/allergy to metoclopramide;
    2. mechanical gastrointestinal obstruction, perforation, or hemorrhage;
    3. seizure disorder;
    4. history of tardive dyskinesia;
    5. or concomitant use of medications/agents likely to increase extrapyramidal reactions.

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2019-09-12 (Actual); Primary Completion 2021-03-10 (Actual); Study Completion 2021-03-10 (Actual)

PRIMARY OUTCOMES:
Change in Brain TSPO availability | One 120-minute PET [11C]PBR28 scan before and one PET [11C]PBR28 scan 2hr after morphine challenge.
  Relative to pre-morphine levels, we will measure the change in brain regional TSPO availability (VT) after morphine. VT will be calculated for brain regions of interest using multi-linear analysis 1 (t*=30) using the metabolite-corrected arterial input function.

SECONDARY OUTCOMES:
Change in Verbal Learning Performance | This Cogstate task will be administered twice: once before and once ~40 minutes after the morphine challenge.
  Relative to pre-morphine levels, we will measure the change in verbal learning performance after morphine via the Cogstate computerized task: International Shopping List. In this task, subjects are asked to memorize and recite (without prompt) 12 common grocery shopping items across 3 trials. Number of correct items recalled across the 3 trials is analyzed.
Change in Verbal Memory Performance | This Cogstate task will be administered twice: once before and once ~70 minutes after the morphine challenge.
  Relative to pre-morphine levels, we will measure the change in verbal memory performance after morphine via the Cogstate computerized task: International Shopping List - Delayed Recall. In this task, subjects are asked to recall (after a time delay) the 12 common grocery shopping items from the International Shopping List task. Number of correct items recalled in this one trial is analyzed.
Change in Psychomotor Speed | This Cogstate task will be administered twice: once before and once ~45 minutes after the morphine challenge.
  Relative to pre-morphine levels, we will measure the change in psychomotor speed via the Cogstate computerized task: Detection. In this task, subjects are asked to respond via button press as soon as the playing card on screen flips over. The log10 of the mean latency to respond (ms) is analyzed.
Change in Visual Attention | This Cogstate task will be administered twice: once before and once ~50 minutes after the morphine challenge.
  Relative to pre-morphine levels, we will measure the change in visual attention via the Cogstate computerized task: Identification. In this task, subjects are asked to respond via button press as soon as he/she identifies that the playing card on screen matches the target card color (red). The log10 of the mean latency to respond (ms) is analyzed.
Change in Visual Learning | This Cogstate task will be administered twice: once before and once ~55 minutes after the morphine challenge.
  Relative to pre-morphine levels, we will measure the change in visual learning via the Cogstate computerized task: One Card Learning. In this task, subjects are asked to respond via button press if he/she identifies that the on-screen playing card has been shown previously. The arc sine of the percent correctly identified is analyzed.
Change in Working Memory (easy) | This Cogstate task will be administered twice: once before and once ~60 minutes after the morphine challenge.
  Relative to pre-morphine levels, we will measure the change in working memory performance via the Cogstate computerized task: One Back. In this task, subjects are asked to respond via button press if he/she identifies that the on-screen playing card matches the card shown just prior to the current card. The log10 of the mean latency to respond (ms) is analyzed.
Change in Working Memory (hard) | This Cogstate task will be administered twice: once before and once ~65 minutes after the morphine challenge.
  Relative to pre-morphine levels, we will measure the change in working memory performance via the Cogstate computerized task: Two Back. In this task, subjects are asked to respond via button press if he/she identifies that the on-screen playing card matches the card shown two prior to the current card. The arc sine of the percent correctly identified is analyzed.
Change in Venous Cytokine/Chemokine Concentration | Plasma samples will be collected 10-minutes before and 60-minutes, 110-minutes, and 250-minutes after the morphine challenge.
  Relative to pre-morphine levels, we will measure the change in venous cytokine and chemokine concentrations (e.g., IL-6, IL-10, TNF-alpha, GM-CSF, and IFN-gamma) periodically after morphine via ELISA assay kit.
Change in Venous Cortisol Concentration | Plasma samples will be collected 10-minutes before and 60-minutes, 110-minutes, and 250-minutes after the morphine challenge.
  Relative to pre-morphine levels, we will measure the change in venous cortisol levels periodically after morphine via ELISA assay kit.
Change in Venous Epinephrine Concentration | Plasma samples will be collected 10-minutes before and 60-minutes, 110-minutes, and 250-minutes after the morphine challenge.
  Relative to pre-morphine levels, we will measure the change in venous epinephrine levels periodically after morphine via ELISA assay kit.
Change in Venous Norepinephrine Concentration | Plasma samples will be collected 10-minutes before and 60-minutes, 110-minutes, and 250-minutes after the morphine challenge.
  Relative to pre-morphine levels, we will measure the change in venous norepinephrine levels periodically after morphine via ELISA assay kit.
Change in Venous Allopregnanolone Concentration | Plasma samples will be collected 10-minutes before and 60-minutes, 110-minutes, and 250-minutes after the morphine challenge.
  Relative to pre-morphine levels, we will measure the change in venous allopregnanolone levels periodically after morphine via ELISA assay kit.
Change in Venous Pregnenolone Concentration | Plasma samples will be collected 10-minutes before and 60-minutes, 110-minutes, and 250-minutes after the morphine challenge.
  Relative to pre-morphine levels, we will measure the change in venous pregnenolone levels periodically after morphine via ELISA assay kit.
Change in Venous Ghrelin Concentration | Plasma samples will be collected 10-minutes before and 60-minutes, 110-minutes, and 250-minutes after the morphine challenge.
  Relative to pre-morphine levels, we will measure the change in venous ghrelin levels periodically after morphine via ELISA assay kit.
Change in Thermal Pain Sensitivity | The Cold Pressor Task will be administered once before and once ~90-minutes after the morphine challenge.
  Relative to pre-morphine levels, we will measure the change in thermal pain sensitivity after morphine via the Cold Pressor Task. Subjects will place their hand in a warm water bath and then a cold water bath. Subjects will be asked to indicate when he/she first experiences pain related to the cold water bath. Time to detection of pain (s) is analyzed.
Change in Thermal Pain Tolerance | The Cold Pressor Task will be administered once before and once ~90-minutes after the morphine challenge.
  Relative to pre-morphine levels, we will measure the change in thermal pain tolerance after morphine via the Cold Pressor Task. Subjects will place their hand in a warm water bath and then a cold water bath. Time to withdrawal his/her hand from the cold water bath (s; max: 90s) is analyzed.
Change in Reward Responsiveness | The Probabilistic Reward Task will be administered once before and once ~260 minutes after morphine.
  Relative to pre-morphine levels, we will measure the change in reward responsiveness after morphine via the computerized Probabilistic Reward Task. Reward responsiveness is calculated as the subject's propensity to modulate his/her response latency to discriminate two stimuli (short and long mouths on a face) based on prior reinforcement (monetary reward for 'correct' responses). This task allows objective measurement of an individuals' responsiveness to monetary reward.

OTHER OUTCOMES:
Change in systolic blood pressure | Blood pressure will be measured 10-minutes before, and 30-minutes, 60-minutes, and 90-minutes after morphine.
  Systolic blood pressure (mmHg; while seated and resting) will be measured periodically before and after morphine.
Change in diastolic blood pressure | Blood pressure will be measured 10-minutes before, and 30-minutes, 60-minutes, and 90-minutes after morphine.
  Diastolic blood pressure (mmHg; while seated and resting) will be measured periodically before and after morphine.
Change in heart rate | Heart rate will be measured 10-minutes before, and 30-minutes, 60-minutes, and 90-minutes after morphine.
  Heart rate (beats per minute; while seated and resting) will be measured periodically before and after morphine.
Change in subjective drug effects | Subjective drug effects measured 10-minutes before, and 30-minutes, 60-minutes, and 90-minutes after morphine.
  Morphine drug effects are measured via visual analogue scale (VAS 0-100mm) for the following adjectives: 'high', 'nauseous', 'good effect', 'bad effect' and 'any effect'.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Woodcock, PhD, Principal Investigator — Yale University; Kelly Cosgrove, PhD, Principal Investigator — Yale University
Locations (1):
- Cosgrove Lab, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant data will be shared upon reasonable request.
Supporting Information: Study Protocol, ICF
Time Frame: Study supporting information will be available upon reasonable request after publication of the primary manuscript.
Access Criteria: Available to research scientists and clinicians for academic uses only.